CLINICAL TRIAL: NCT01867203
Title: Lipid-lowering Therapy Individualization
Brief Title: Functional and Clinical Impact of CYP3A Genetic Polymorphisms on Statin Therapy
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: CYPstatin001
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Patients With High Cholesterol Levels Needing a Lipid-lowering Therapy
MeSH Terms: interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Statin users
  Interventions: Other: Genotyping

INTERVENTIONS:
Other: Genotyping — DNA extraction from blood

SUMMARY:
Patients needing lipid lowering therapy will be recruited before initiation of the treatment. For each patient, total and LDL cholesterol levels before start of therapy will be measured. One, three and six months after his/her first visit, when steady-state will be reached, for each included patient, the cholesterol levels will be re-assessed in order to evaluate the response to statin therapy calculated as the amplitude of cholesterol reduction. The aim is to assess the association between patient's genotype and the response to statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient known to be compliant
* Age [25-80]
* treated with Atorvastatin, simvastatin, fluvastatin.

Exclusion Criteria:

* Pregnancy

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with statin drugs
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Cholesterol levels-side effects | 1 to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Luc Hospital, Brussels, Belgium